CLINICAL TRIAL: NCT00785460
Title: Benfotiamine Prevents Vascular Dysfunction in Healthy Smokers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Alin Stirban, Heart and Diabetes Center NRW
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Benfo Smoker
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Last update posted 2008-11-05 (Estimated); Status verified 2008-11

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — benphothiamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Benfotiamine and Smoking (Experimental)
  Interventions: Drug: Benfotiamine
- Smoking alone (Placebo Comparator)
  Interventions: Drug: Benfotiamine

INTERVENTIONS:
Drug: Benfotiamine

SUMMARY:
Benfotiamine pretreatment (3 days)at high dosage (1050 mg/day) prevents in healthy subjects smoking-induced vascular dysfunction assessed by ultrasound flow mediated dilatation of the brachial artery.

DETAILED DESCRIPTION:
Benfotiamine pretreatment (3 days)at high dosage (1050 mg/day) prevents in healthy subjects smoking-induced vascular dysfunction assessed by ultrasound flow mediated dilatation (FMD) of the brachial arteryand laboratory parameters (adhesion molecules).

ELIGIBILITY:
Inclusion Criteria:

* healthy habitual smokers

Exclusion Criteria:

* any kind of chronic disease

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-01; Primary Completion 2008-05

PRIMARY OUTCOMES:
Flow mediated dilatation | 3 days

SECONDARY OUTCOMES:
Laboratory markers of endothelial function | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Alin Stirban, MD, Principal Investigator — Ruhr-University Bochum
Locations (1):
- Heart and Diabetes Center, Bad Oeynhausen, North Rhine-Westphalia, Germany